CLINICAL TRIAL: NCT04986956
Title: Longitudinal Study to Assess the Effects of Whole Coffee Cherry Extract (WCCE)
Brief Title: Whole Coffee Cherry Study
Acronym: WCCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: VDF FutureCeuticals Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer L. Robinson, Ph.D., Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: #21-219
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Effect of Drug
Keywords: coffee cherry; cognition; virtual study; internet

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups - study materials (whole coffee cherry extract (WCCE) or placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding information will be held by the study sponsor, VDF FutureCeuticals, Inc. The study will be conducted in a double-blind fashion such that both the investigators and the participants are unaware of their assignment. Unblinding will only occur once the study has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo will be a simple microcellulose, which is generally-recognized-as-safe (GRAS) and commonly used in food products.
  Interventions: Dietary Supplement: Placebo
- Whole coffee cherry extract (Active Comparator): Whole coffee cherry extract (WCCE; otherwise known as the generally-recognized-as-safe (GRAS) supplement Neurofactor(TM)), is a proprietary, safe, powdered extract of whole coffee cherries from coffea arabica with high levels of polyphenols and substantially low (<2%; <4mg) levels of caffeine. The only content of the supplement is WCCE - there are no excipients, binders, or flow agents, nor are there any other materials. The coffee cherry is subjected to a food-grade water ethanol extraction; thus, after extraction, only 100% coffee-based components remain. 200mg of WCCE will be administered daily for 28 days.
  Interventions: Dietary Supplement: Whole coffee cherry extract

INTERVENTIONS:
Dietary Supplement: Whole coffee cherry extract — 200mg WCCE
  Other Names: WCCE; CCE
  Arms: Whole coffee cherry extract
Dietary Supplement: Placebo — Placebo for comparison to WCCE
  Arms: Placebo

SUMMARY:
There has been increasing interest in natural dietary supplements that may support healthy cognition. Recent studies have demonstrated promising effects of bioactive phytochemicals (e.g., polyphenols) on cardiovascular and endocrine health outcomes. As such, an increasingly intriguing line of inquiry is whether materials high in these compounds may also have effects on psychological measures. Preliminary evidence suggests that polyphenols may improve cognition, for example, particularly in aging populations. Whole coffee cherry extract (WCCE; otherwise known as the generally-recognized-as-safe (GRAS) supplement Neurofactor(TM)), is a proprietary, safe, powdered extract of whole coffee cherries from coffea arabica with high levels of polyphenols and substantially low (<2%; <4mg) levels of caffeine. WCCE has been previously associated with increased serum concentrations of both circulating and exosomal brain derived neurotrophic factor (BDNF), in addition to increased alertness and decreased fatigue. However, few well-powered and well-designed studies have been conducted despite the mounting preliminary evidence. Here, the investigators propose a study to examine the long-term effects of a 200mg dose of WCCE on measures of cognition.

DETAILED DESCRIPTION:
The investigators will conduct a virtual study whereby participants will be given either 200mg WCCE or placebo to take every day for 28 days. Every 7 days, participants will take a cognitive assessment via the internet using a platform called Millisecond (https://www.millisecond.com/). The cognitive assessment will be composed of tasks that broadly test working memory, focus, and attention. Compliance checks will be administered daily via the participant's smartphone. This study will be conducted in a double-blind fashion, such that the experimental team and the participants are unaware of group assignment (200mg vs. placebo). Blinding information will be held by the study sponsor, VDF FutureCeuticals, Inc. Group assignment will be determined by random number generator, with restrictions to ensure equal group sizes, and equal distribution of males/females in each group. Participants, between 40-65 years of age, with no known psychiatric or neurological conditions, will be recruited from the general community via online advertisements, social media posts, community flyers, and newspaper ads (if needed). Participants will be excluded if they are taking medications known to alter cognitive functioning (psychotropic medications such as fluoxetine, benzodiazepines, etc. or other medications such as insulin). The primary variables of interest will be the behavioral performance on the cognitive tasks over time, inclusive of reaction time and accuracy. Compensation will be commensurate with study participation, with a maximum payout of $125.

ELIGIBILITY:
Inclusion Criteria:

* Between 40-65 years of age
* No diagnosed psychiatric or neurological condition
* Reliable internet service
* Moderate computer literacy
* Individuals must have a smartphone
* Individuals must have a laptop, desktop, or iPad

Exclusion Criteria:

* Individuals taking medications known to alter cognitive functioning (e.g., psychotropic medications such as fluoxetine, benzodiazepines, etc.)
* Individuals taking medications that alter metabolic function, such as insulin or metformin.
* Shift workers
* Health conditions that would prevent an individual from successfully completing the study (I.e., motor control conditions such as Parkinson's, or psychiatric conditions such as ADHD)
* Individuals with metabolic conditions
* Have had or currently have cancer
* Have taken CBD or multivitamins in the last 2 weeks
* Individuals with unreliable or no internet access/service
* Individuals who are unable to use a smartphone or are lacking the computer literacy necessary to complete the study remotely
* Individuals without a laptop, desktop or iPad that would prevent them from completing the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Behavioral Measures - Change in Go/NoGo Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in N-back Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction/accuracy time for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Face-Name Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Stroop Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Flanker Task Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Symbol Search Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Trail Making Reaction Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Face in the Crowd Time | Collected at baseline (pre- and post-consumption) and then once weekly (pre-consumption) through the duration of the study (approximately 28 days)
  Response/reaction time/accuracy for each stimuli will be recorded in ms using Inquisit. Reaction times will be calculated for correct and incorrect trials separately.

SECONDARY OUTCOMES:
Daily Self-reported Sleep | The question will be administered daily for the duration of the study (approximately 28 days)
  The investigators will assess changes in the amount of sleep a participant had on a daily basis for the entire duration of the study via a single daily question asking about the number of hours of sleep the participant had the night before.
Weekly Self-reported Sleep Hygiene | Questions are administered weekly for the duration of the study (approximately 28 days)
  The investigators will assess changes in sleep via an in-house questionnaire (administered every 7 days for the entire length of the study) that inquires about the quality of sleep for the past 7 days, as well as how the participant would rate their sleep for the night prior to the assessment. These questions are scored as 1 = excellent, 2 = good, 3 = average, 4 = poor, and 5 = terrible.
Weekly Self-reported Mood | The questionnaire is administered weekly for the duration of the study (approximately 28 days)
  The investigators will assess changes in mood every 7 days for the duration of the study. This questionnaire, developed in-house, asks about how often the participant has felt alert, focused, attentive, in-control, sleepy, determined, motivated, happy, and upset the participant has felt in the last 7 days. The scale is scored as 1 = always, 2 = most of the time, 3 = about half of the time, 4 = sometimes, and 5 = never.
Daily Self-reported Mood | The question will be administered daily for the duration of the study (approximately 28 days)
  The investigators will assess changes in mood via a daily question about how good/bad the participant feels on a scale of 0-100 (0 being worst they have ever felt, and 100 being the best they have ever felt).

OTHER OUTCOMES:
Compliance | Daily for the duration of the study (approximately 28 days)
  The investigators will assess compliance via daily questionnaires delivered to the participant's smartphone.

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao H, Ou J, Chen L, Zhang Y, Szkudelski T, Delmas D, Daglia M, Xiao J. Dietary polyphenols and type 2 diabetes: Human Study and Clinical Trial. Crit Rev Food Sci Nutr. 2019;59(20):3371-3379. doi: 10.1080/10408398.2018.1492900. Epub 2018 Nov 19. PMID 29993262
- [Background] Hurtado-Barroso S, Quifer-Rada P, Rinaldi de Alvarenga JF, Perez-Fernandez S, Tresserra-Rimbau A, Lamuela-Raventos RM. Changing to a Low-Polyphenol Diet Alters Vascular Biomarkers in Healthy Men after Only Two Weeks. Nutrients. 2018 Nov 14;10(11):1766. doi: 10.3390/nu10111766. PMID 30441880
- [Background] Mendonca RD, Carvalho NC, Martin-Moreno JM, Pimenta AM, Lopes ACS, Gea A, Martinez-Gonzalez MA, Bes-Rastrollo M. Total polyphenol intake, polyphenol subtypes and incidence of cardiovascular disease: The SUN cohort study. Nutr Metab Cardiovasc Dis. 2019 Jan;29(1):69-78. doi: 10.1016/j.numecd.2018.09.012. Epub 2018 Oct 4. PMID 30459074
- [Background] Schuster J, Mitchell ES. More than just caffeine: psychopharmacology of methylxanthine interactions with plant-derived phytochemicals. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:263-274. doi: 10.1016/j.pnpbp.2018.09.005. Epub 2018 Sep 10. PMID 30213684
- [Background] Sarubbo F, Moranta D, Pani G. Dietary polyphenols and neurogenesis: Molecular interactions and implication for brain ageing and cognition. Neurosci Biobehav Rev. 2018 Jul;90:456-470. doi: 10.1016/j.neubiorev.2018.05.011. Epub 2018 May 23. PMID 29753753
- [Background] Shukitt-Hale B, Miller MG, Chu YF, Lyle BJ, Joseph JA. Coffee, but not caffeine, has positive effects on cognition and psychomotor behavior in aging. Age (Dordr). 2013 Dec;35(6):2183-92. doi: 10.1007/s11357-012-9509-4. Epub 2013 Jan 24. PMID 23344884
- [Background] Whyte AR, Cheng N, Fromentin E, Williams CM. A Randomized, Double-Blinded, Placebo-Controlled Study to Compare the Safety and Efficacy of Low Dose Enhanced Wild Blueberry Powder and Wild Blueberry Extract (ThinkBlue) in Maintenance of Episodic and Working Memory in Older Adults. Nutrients. 2018 May 23;10(6):660. doi: 10.3390/nu10060660. PMID 29882843
- [Background] Robinson JL, Hunter JM, Reyes-Izquierdo T, Argumedo R, Brizuela-Bastien J, Keller R, Pietrzkowski ZJ. Cognitive short- and long-term effects of coffee cherry extract in older adults with mild cognitive decline. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2020 Nov;27(6):918-934. doi: 10.1080/13825585.2019.1702622. Epub 2019 Dec 12. PMID 31829793
- [Background] Robinson JL, Yanes JA, Reid MA, Murphy JE, Busler JN, Mumford PW, Young KC, Pietrzkowski ZJ, Nemzer BV, Hunter JM, Beck DT. Neurophysiological Effects of Whole Coffee Cherry Extract in Older Adults with Subjective Cognitive Impairment: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Pilot Study. Antioxidants (Basel). 2021 Jan 20;10(2):144. doi: 10.3390/antiox10020144. PMID 33498314
- [Background] Heimbach JT, Marone PA, Hunter JM, Nemzer BV, Stanley SM, Kennepohl E. Safety studies on products from whole coffee fruit. Food Chem Toxicol. 2010 Aug-Sep;48(8-9):2517-25. doi: 10.1016/j.fct.2010.06.025. Epub 2010 Jun 18. PMID 20600539
- [Background] Yashin A, Yashin Y, Wang JY, Nemzer B. Antioxidant and Antiradical Activity of Coffee. Antioxidants (Basel). 2013 Oct 15;2(4):230-45. doi: 10.3390/antiox2040230. PMID 26784461
- [Background] Reed, R.A., et al., Acute Low and Moderate Doses of a Caffeine-Free Polyphenol-Rich Coffeeberry Extract Improve Feelings of Alertness and Fatigue Resulting from the Performance of Fatiguing Cognitive Tasks. Journal of Cognitive Enhancement, 2018.
- [Background] Reyes-Izquierdo T, Nemzer B, Shu C, Huynh L, Argumedo R, Keller R, Pietrzkowski Z. Modulatory effect of coffee fruit extract on plasma levels of brain-derived neurotrophic factor in healthy subjects. Br J Nutr. 2013 Aug 28;110(3):420-5. doi: 10.1017/S0007114512005338. Epub 2013 Jan 14. PMID 23312069
- [Background] Abdel-Aziz K, Larner AJ. Six-item cognitive impairment test (6CIT): pragmatic diagnostic accuracy study for dementia and MCI. Int Psychogeriatr. 2015 Jun;27(6):991-7. doi: 10.1017/S1041610214002932. Epub 2015 Jan 29. PMID 25630996